CLINICAL TRIAL: NCT04467138
Title: High Dose Intravenous Fish Oil Reduces Inflammation and Improves Liver Function
Brief Title: High Dose Intravenous Fish Oil Reduces Inflammation
Status: Completed | Type: Observational
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Unit, Stanley Dudrick's Memorial Hospital
Other Study IDs: Omegaven
Record Dates: First submitted 2020-07-05; First posted 2020-07-10 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Lipid Metabolism Disorders
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — fish oil triglycerides; Fish Oils

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory bowel disease: Patients with either Crohn's disease (CD, n=22), and Ulcerative colitis (UC, n=19).
  Interventions: Drug: Omegaven
- Chronic intestinal failure: Patients with intestinal failure (CIF, n=20)
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Pure fish oil emulsion (Omegaven®, Fresenius Kabi) was used as the additional product along with the standard lipid emulsion to reach a fish oil dose of approx. 0.5 g fish oil/kg/d.
  Other Names: Fish oil

SUMMARY:
Retrospective analysis of 51 patients (27 female, 24 male, mean age 51.5±12.6 years) who received all-in-one PN including amino acids, glucose and lipids supplemented with pure fish oil LE was performed.

DETAILED DESCRIPTION:
All patients depended on parenteral nutrition (PN) are prone to inflammation. This condition may aggravate already existing proinflammatory status and can become a critical factor for developing liver dysfunction (LD). Intravenous fish oil may attenuate the inflammatory status, , however, data on its use in adults is scarce. The aim of the study was to investigate the impact of the addition of pure fish oil intravenous lipid emulsion (ILE) as part of short- and long term PN in patients either at risk or with already existing inflammation.

Retrospective analysis of 51 patients (27 female, 24 male, mean age 51.5±12.6 years) who received all-in-one PN including amino acids, glucose and lipids supplemented with pure fish oil LE was performed. Pure fish oil emulsion (Omegaven®, Fresenius Kabi) was used as the additional product along with the standard lipid emulsion to reach a fish oil dose of approx. 0.5 g fish oil/kg/d. Diagnoses were chronic intestinal failure (CIF, n=20), Crohn's disease (CD, n=22), and Ulcerative colitis (UC, n=19). The observation period was 12 months for CIF and 21days for UC and CD.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age,
* metabolic stability (the absence of pathological laboratory resulting in the change of PN regime for at least one month)
* ability to tolerate up to 1.0 g lipids/kg body weight per day as a part of PN.

Exclusion Criteria:

* patients with a history of cancer and anti-cancer treatment within the last 5 years, severe hyperlipidemia, severe coagulopathy, severe renal insufficiency, acute thromboembolic events, positive test for HIV, Hepatitis B or C (from medical history), known or suspected drug or alcohol abuse, participation in another interventional clinical trial in parallel or within three months prior to the start of this clinical trial, for women with childbearing potential (i.e. females who are not chemically or surgically sterile or females who are not postmenopausal) or women of childbearing potential tested positive on standard pregnancy test (urine dipstick) or/and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either inflammatory bowel disease or chronic intestinal failure. Both in and out patients
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in hsCRP concentration | 4 weeks
  Serum concentration of hsCRP (pg/mL)
Change in Il-6 concentration | 4 weeks
  Serum concentration of Il-6 (pg/mL)
Change in interleukin-10 concentration | 4 weeks
  Serum concentration of IL-10 (pg/mL)
Change in procalcytonin concentration | 4 weeks
  Serum concentration of procalcytonin (ng/mL)
Change in bilirubin concentration | 4 weeks
  Serum concentration of bilirubin (umol/L)
Change in SGPT concentration | 4 weeks
  Serum concentration of SGPT(U/l)
Change in SGOT concentration | 4 weeks
  Serum concentration of SGOT (U/l)
Change in alkaline phosphatase concentration | 4 weeks
  Serum concentration of alkaline phosphatase (U/l)
Change in C-reactive protein concentration | 4 weeks
  Serum concentration of CRP (mg/l)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, PhD, Principal Investigator — 1972
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klek S, Szczepanek K, Scislo L, Walewska E, Pietka M, Pisarska M, Pedziwiatr M. Intravenous lipid emulsions and liver function in adult chronic intestinal failure patients: results from a randomized clinical trial. Nutrition. 2018 Nov;55-56:45-50. doi: 10.1016/j.nut.2018.03.008. Epub 2018 Mar 22. PMID 29960156